CLINICAL TRIAL: NCT00315640
Title: A Study of the Safety and Efficacy of Anecortave Acetate for Treatment of Steroid Induced Intraocular Pressure (IOP) Elevation
Brief Title: Anecortave Acetate for Treatment of Steroid Induced Intraocular Pressure (IOP) Elevation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-05-03; 2005-001598-93
Record Dates: First submitted 2006-04-17; First posted 2006-04-19 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2010-01

CONDITIONS: Eye Diseases
Keywords: Elevated IOP due to intravitreal triamcinolone therapy
MeSH Terms: conditions — Eye Diseases | interventions — anecortave acetate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Anecortave Acetate 3 mg Depot (Experimental): One 0.5 mL anterior juxtascleral depot (AJD) injection in the study eye
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 6 mg/mL
- Anecortave Acetate 15 mg Depot (Experimental): One 0.5 mL anterior juxtascleral depot (AJD) injection in the study eye
  Interventions: Drug: Anecortave Acetate Suspension Depot, 30 mg/mL
- Anecortave Acetate 30 mg Depot (Experimental): One 0.5 mL anterior juxtascleral depot (AJD) injection in the study eye
  Interventions: Drug: Anecortave Acetate Sterile Suspension, 60 mg/mL
- Anecortave Acetate Vehicle (Other)
  Interventions: Other: Anecortave Acetate Vehicle

INTERVENTIONS:
Drug: Anecortave Acetate Sterile Suspension, 6 mg/mL — One 0.5 mL anterior juxtascleral depot (AJD) injection in the study eye
  Arms: Anecortave Acetate 3 mg Depot
Drug: Anecortave Acetate Suspension Depot, 30 mg/mL — One 0.5 mL anterior juxtascleral depot (AJD) injection in the study eye
  Arms: Anecortave Acetate 15 mg Depot
Drug: Anecortave Acetate Sterile Suspension, 60 mg/mL — One 0.5 mL anterior juxtascleral depot (AJD) injection in the study eye
  Arms: Anecortave Acetate 30 mg Depot
Other: Anecortave Acetate Vehicle — One 0.5 mL anterior juxtascleral depot (AJD) injection in the study eye
  Arms: Anecortave Acetate Vehicle

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of anecortave acetate depot when administered for the treatment of elevated IOP following treatment with steroids.

ELIGIBILITY:
Inclusion Criteria:

* Either gender
* 18 years of age or older
* IOP elevation caused by steroid usage
* Other protocol-defined inclusion criteria may apply

Exclusion Criteria:

* Under 18 years of age
* Other protocol-defined exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2005-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Mean change in IOP at Week 4 from Baseline | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Landry, Study Director — Alcon Research
Locations (12):
- United States (5):
  - Jacksonville, Jacksonville, Florida
  - Miami, Miami, Florida
  - Detroit, Detroit, Michigan
  - Fort Worth, Texas
  - Houston, Houston, Texas
- San Paulo, São Paulo, Brazil
- Budapest, Budapest, Hungary
- Padova, Padua, Italy
- Amsterdam, Amsterdam, Netherlands
- Bayamon, Bayamón, Puerto Rico
- Barcelona, Barcelona, Spain
- Newcastle upon Tyne, Newcastle upon Tyne, United Kingdom